CLINICAL TRIAL: NCT02604693
Title: Exposure in Epigenetic Regulation of Immune Response in Chronic Beryllium
Brief Title: Exposure in Epigenetic Regulation of Immune Response in Chronic Beryllium Disease (CBD)
Acronym: BeEpiGen
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Lisa Maier, MD, National Jewish Health
Other Study IDs: HS-2866
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Chronic Beryllium Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chronic Beryllium Disease: Those that have been diagnosed with the disease. No interventions will be administered.
  Interventions: Other: Nothing
- Beryllium Sensitization: Those that have been diagnosed with beryllium sensitization and do not have chronic beryllium disease. No interventions will be administered.
  Interventions: Other: Nothing
- normal controls: Those that do not have chronic beryllium disease or beryllium sensitization. No interventions will be administered
  Interventions: Other: Nothing

INTERVENTIONS:
Other: Nothing — No interventions will be administered.

SUMMARY:
This study will provide important results for each aim, while also providing an integrative transcriptional and epigenomic profile of CBD.

In Aim 1 the Investigator will define genome-wide epigenetic alterations of CBD, by determining genes that are DM in pivotal immune cells, in the target organ (CD4+ BAL cells) in CBD compared to BeS and healthy controls. In addition, the Investigator will determine the impact of Be exposure on the methylation profile of CBD and BeS cells compared to each other and normal controls. This information will be used to define DM regions, genes and their networks.

Using the cases and controls from Aim 1, we will evaluate the gene-expression from these same subjects in Aim 2 to define functional epigenetic loci based on DE in CD4+ BAL cells with and without Be exposure. The Investigator will also integrate ENCODE/RE methylation, histone modification, and chromatin accessibility data as well as our genome-wide association study (GWAS) data to prioritize epigenetic marks and networks for confirmation and validation in Aim 3. In Aim 3, the Investigator will test the generalizability of their findings, explore the potential of methylation marks as biomarkers of disease in PBMCs and determine if change in methylation of these targets with AZA or folic acid affects key immune and regulatory pathways in a second set of CBD and BeS subjects. Throughout the Aims, the Investigator will use both fresh CD4+ T cells to directly assess disease relevance and Be-stimulated cultured CD4+ T cells (compared to unstimulated cultured T cells) to assess the impact of environmental exposure .

ELIGIBILITY:
Inclusion Criteria:

Chronic Beryllium Disease (CBD):

1. History of Beryllium exposure
2. Positive blood and/or bronchoalveolar lavage (BAL) Beryllium Lymphocyte Proliferation Tests (BeLPT)
3. Biopsy-proven pathologic changes consistent with CBD, specifically non-caseating granulomas and/or mononuclear cell interstitial infiltrates.

Beryllium Sensitization:

1. History of Beryllium exposure
2. Two or more positive blood beryllium lymphocyte proliferation tests (BeLPT) or positive bronchoalveolar lavage (BAL) BeLPT
3. Normal lung tissue (no histology suggestive of CBD).

Normal Controls:

1. No history of beryllium exposure
2. Former smokers or never smokers -

Exclusion Criteria:

Chronic Beryllium Disease:

1. Immunosuppressive therapy within the last three months
2. Current cigarette smoking or smoking within six months prior to the study
3. Positive lung washing or biopsy cultures for fungi, mycobacteria or other respiratory pathogen consistent with an acute or chronic infection
4. Weight less than 110 lbs. (for venipuncture)
5. Pregnancy
6. Severe room air hypoxemia and or hypercapnia (precluding BAL), e.g., resting PaO2 < 45, PaCO2 > 45 mm Hg; (Denver altitude 5,280 feet)
7. Presence of another disease that may be expected to significantly affect patient mortality and or the immune response (e.g., HIV, HCV, cancer, uncorrected bleeding diathesis, acute hypercapnia with a resting PaCO2 above 45 mm Hg; serious cardiac arrhythmia, recent myocardial infarction within 6 weeks)
8. Patient inability to participate in the study, such as inability to undergo venipuncture and BAL procedures that form part of the inclusion/exclusion criteria or part of the outcome measure

Beryllium Sensitization:

1. Known underlying systemic or lung disease;
2. Current cigarette smoking or smoking within six months prior to the study
3. Positive lung pathology consistent with CBD
4. Pregnancy
5. Weight less than 110 lbs. (for venipuncture)
6. Presence of another disease that may be expected to significantly affect patient mortality and or the immune response (e.g., HIV, HCV, cancer, uncorrected bleeding diathesis, serious cardiac arrhythmia; recent myocardial infarction within 6 weeks)
7. Patient inability to participate in the study, such as inability to undergo venipuncture and BAL procedures that form part of the inclusion/exclusion criteria or part of the outcome measure

Normal Controls:

1. History of beryllium exposure
2. Known underlying systemic or lung disease;
3. Immunosuppressive therapy or other medication for as systemic disease process in the last 3 months;
4. Current smokers or smoking within 6 months of study
5. Pregnancy
6. Weight less than 110 lbs. (for venipuncture)
7. Inability to undergo BAL or venipuncture procedures -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll subjects using standard case and control definitions. We will enroll up to 150 subjects. Controls will be frequency matched on age, gender, race and smoking status to limit methylation changes related to these factors.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2014-12-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Determine the critical immune and environmentally-induced epigenetic alterations in the CD4+ T cells at the site of disease involvement from CBD compared to BeS and control subjects. | Year 1 through year 2
  The Investigators goal is to define an epigenomic profile for BeS and CBD and for Be exposure in the lung. Most studies using similar methods have demonstrated significant hypo- and hyper-methylation, in disease states, which we also expect to find. In addition, we expect to confirm an association between CBD and Th1 epigenetic regulation, finding DM in regions such as FOXP3, Th1 differentiation pathways and TNFalpha, likely with modulation of these and other regions with Be exposure. There is no information regarding methylation alterations induced by an immune mediated exposure such as Be. The investigator expects to define new and unique genes with DM, some involved in the immune response and others in pathways and networks not known to be associated with granulomatous inflammation, shedding light on the pathogenesis of this and similar diseases.
Define the functional impact of critical immune and environmentally-induced epigenetic alterations in gene expression from BAL CD4+ T cells from CBD compared to BeS and control subjects used in Aim 1 | year 1 through year 4
  At the end of Aim 2, the Investigator will have 20 genes with validated methylation and expression changes. These methylation changes are likely to be regulatory in CD4+ T cells not only based on relationship with expression but also network analysis of methylation changes (Aim 1), relationship with immune cell phenotypes, cell specific chromatin/histone marks from ENCODE and RE datasets, and our CBD GWAS SNPs (Aim 2). The Investigator has a pipeline of data analysis currently in place as evidenced by our preliminary data; as new approaches such as these become available, we will use them to analyze our data.

SECONDARY OUTCOMES:
Test the generalizability of our findings and validity of identified methylation and gene expression changes as potential biomarkers and therapeutic targets. | Year 3 through year 5
  This Aim will result in a set of key data, including potential new biomarkers of disease and exposure in CBD. The Investigator expects to be able to validate the 20 loci identified in Aim 2 in BAL as well as PBMCs. Even with a sample size of n=10 in their gene-expression studies, the Investigator was able to define significant DE in PBMCs in CBD that they are currently exploring as biomarkers in a larger population; the Investigator expects that with changes found evaluating the relationship between DM and DE that they will be able to use the PBMCs as a biomarker of disease and exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Maier, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States